CLINICAL TRIAL: NCT06914245
Title: Towards Personalized Care Pathways for Bowel Symptoms in Rectal Cancer Patients Through Precision Medicine
Brief Title: Personalized Care Pathways for Bowel Symptoms in Rectal Cancer Patients_contributing Factors (Treatable)
Acronym: Treatable
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: AZ Delta (Other); Universitair Ziekenhuis Brussel (Other); Ziekenhuis aan de Stroom (Other); AZ Oostende (Unknown); General Hospital Groeninge (Other); Heilig Hart Ziekenhuis Lier (Unknown); Meander MC, Amersfoort, the Netherlands (Unknown); AZORG (Unknown); UZ Leuven, Leuven, Belgium (Unknown)
Responsible Party: Principal Investigator, Inge Geraerts, Professor Dr., KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S69283
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; LARS - Low Anterior Resection Syndrome; Active Surveillance
Keywords: Bowel diary; Quality of Life (QoL); Care pathway
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TME/PME (Experimental): To investigate the prognostic variables of persistent bowel symptoms and persistent consequences of bowel symptoms, specifically the impact on QoL, participants scheduled for rectal surgery will be asked to complete an electronic bowel diary on their mobile phones and to fill out several online questionnaires at multiple time points (prior to surgery, and at 1, 6, and 12 months post-rectal surgery or post-stoma closure).
  Interventions: Diagnostic Test: Electronic bowel diary; Diagnostic Test: Faecal Incontinence Quality of Life questionnaire (FIQL); Diagnostic Test: EuroQoL 5 dimensions, 5 levels (EQ-5D-5L)
- Active surveillance (Experimental): To investigate the prognostic variables of persistent bowel symptoms and persistent consequences of bowel symptoms, specifically the impact on QoL, participants in active surveillance will be asked to complete an electronic bowel diary on their mobile phones and to fill out several online questionnaires at multiple time points (at baseline and at 1, 6, and 12 months after completion of neoadjuvant therapy).
  Interventions: Diagnostic Test: Electronic bowel diary; Diagnostic Test: Faecal Incontinence Quality of Life questionnaire (FIQL); Diagnostic Test: EuroQoL 5 dimensions, 5 levels (EQ-5D-5L)

INTERVENTIONS:
Diagnostic Test: Electronic bowel diary — This bowel diary will be available on the smartphone in the form of an application.
Diagnostic Test: Faecal Incontinence Quality of Life questionnaire (FIQL) — This questionnaire will be available online.
Diagnostic Test: EuroQoL 5 dimensions, 5 levels (EQ-5D-5L) — This questionnaire will be available online.

SUMMARY:
Colorectal cancer is the 2nd and 3rd most common cancer in respectively women and men, of which about 40% is located in the rectum. The gold standard treatment for rectal cancer (RC) is a low anterior resection combined with chemoradiotherapy. However, this treatment negatively affects various aspects of bowel function and patients' quality of life. These bowel symptoms often remain prevalent, even 12 months after RC treatment.

The aim of this study is to identify the factors contributing to persistent bowel symptoms and their long-term impact on quality of life following treatment for rectal cancer, assessed 12 months after surgery or stoma closure in surgically treated patients, and 12 months after completion of neoadjuvant therapy in patients managed with active surveillance/watch-and-wait. These insights are crucial for developing an effective care approach, as they help determine when specific evaluations should be conducted and which treatments should be applied at different stages.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
* At least 18 years of age at the time of signing the Informed Consent Form (ICF).
* Proficient in reading, comprehending, and conversing in Dutch.
* Patients scheduled for Total Mesorectal Excision (TME) or Partial Mesorectal Excision (PME) or 'Watch and wait' protocol due to rectal cancer.

Exclusion Criteria:

* The participant has undergone a different type of surgery, including a Hartmann procedure, abdominoperineal excision, transanal endoscopic microsurgery, or sigmoid resection.
* Experienced fecal incontinence prior to undergoing surgery.
* Are affected by neurological disorders affecting bowel function.
* Already underwent previous pelvic radiation or rectal surgery for non-cancer reasons.
* Has a permanent stoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Bowel symptoms after rectal cancer treatment | 12 months
  To ensure that patients can report all their bowel symptoms where they suffer from, a valid, reliable, user-friendly, and easy-to-interpret electronic bowel diary has been developed in another research project for which approval has already been obtained from the Ethical Committee of the University Hospitals Leuven (S68746). This electronic bowel diary will be used to map out all bowel complaints.
The evaluation of Quality of Life (QoL) related to bowel symptoms after rectal cancer treatment | 12 months
  Faecal Incontinence Quality of Life questionnaire (FIQL) will be used for the evaluation of QoL related to faecal incontinence problems. The FIQL is a reliable and valid 41-item questionnaire, resulting in 4 subscales: Lifestyle, Coping/behavior, Depression/Self Perception and Embarrassment. The Scales ranges from 1 to 5, with a 1 indicating a lower functional status of quality of life. This questionnaire is also validated in Dutch.
The evaluation of overall Quality of Life (QoL) after rectal cancer treatment | 12 months
  EuroQol 5 Dimensions, 5 Levels (EQ-5D-5L) will be used to assess overall quality of life (QoL). The EQ-5D-5L is a reliable and valid 6-item questionnaire, consisting of two parts: the social perspective and the individual perspective of one's own health.
  In the social perspective, the health state is converted into a value set with a score ranging from 0 to 1, where 0 represents being dead and 1 represents full health. The individual perspective assesses the respondent's own perception of their health, with a score ranging from 0 to 100.
  This questionnaire is validated in Dutch and widely used to measure general health-related quality of life.

SECONDARY OUTCOMES:
The predictive value of 'defecation functions' measured with the MSKCC-BFI for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Defecation functions will be assessed with the Memorial Sloan-Kettering Cancer Centre Bowel Function Instrument (MSKCC-BFI). The MSKCC-BFI is a broad bowel specific questionnaire (18 items), resulting in three subscales, four single items and one total score for bowel function.
The predictive value of 'defecation functions' measured with the LARS score for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Defecation functions will be assessed with the LARS score. The LARS score is a short questionnaire, consisting of 5 items, stratifying patients into no, minor or major LARS. This questionnaire has been validated in Dutch.
The predictive value of 'defecation functions' measured with the PAC-SYM for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Defecation functions will be assessed with the Patient Assessment of Constipation-Symptoms questionnaire (PAC-SYM). The PAC-SYM is a validated constipation-specific questionnaire of 12 items that reflect stool, rectal and abdominal symptoms. Patients report the severity of each symptom on a Likert scale from 0 (absent) to 4 (very severe). This questionnaire has been validated in Dutch.
The predictive value of 'baseline age' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | pre-operatively, prior to the surgical intervention for rectal cancer
  Information concerning the patient age will be derived from the medical file.
The predictive value of 'gender' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | pre-operatively, prior to the surgical intervention for rectal cancer
  Information concerning the gender of the patient will be derived from the medical file.
The predictive value of 'diabetes' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | pre-operatively, prior to the surgical intervention for rectal cancer
  Information concerning diabetes will be derived from the medical file.
The predictive value of 'smoking history' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | pre-operatively, prior to the surgical intervention for rectal cancer
  Information concerning smoking history (current, former, never) will be queried.
The predictive value of 'BMI' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | pre-operatively, prior to the surgical intervention for rectal cancer
  Information regarding the patient's BMI will be collected pre-operatively.
The predictive value of 'depression' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Depression will be measured using the Patient Health Questionnaire (PHQ-9), a 9-item validated Dutch questionnaire with scores ranging from 0 to 27.
  Higher scores indicate more severe depression, classifying patients into mild, moderate, moderately severe, or severe depression.
The predictive value of 'anxiety' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Anxiety will be assessed using the Generalized Anxiety Disorder-7 (GAD-7), a 7-item validated Dutch questionnaire with a score range of 0 to 21. Higher scores reflect greater anxiety severity, categorizing patients into mild, moderate, or severe anxiety.
The predictive value of 'resilience' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | 12 months
  Resilience will be measured using the Connor-Davidson Resilience Scale (CD-RISC), a 10-item questionnaire with scores ranging from 0 to 40, where higher scores indicate greater resilience. The scale was translated into Dutch using the forward-backward translation technique to ensure accuracy.
The predictive value of 'Optimal physiotherapy care' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | at 6 months post-surgery or post-stoma closure
  The assessment of optimal physiotherapy care for bowel symptoms during and after RC treatment will be defined based on available scientific evidence, guidelines and clinical expertise of the promotors of this project. Through a self-developed questionnaire, patients will be questioned which care they received in order to estimate by the research team whether they received no/suboptimal/optimal PT care.
The predictive value of 'Treatment-related factors' for the development of persistent bowel symptoms and consequences of bowel symptoms at 12 months post-surgery or post-stoma closure | At 1 month post-surgery or post-stoma closure
  TNM-stage, tumor height, neoadjuvant therapy, stoma prior to surgery, date rectal cancer surgery, approach rectal resection, surgery technique, reconstruction technique, type of anastomosis, Rullier classification, inferior mesenteric artery ligation, inferior mesenteric vein ligation, type of stoma, date stoma closure, adjuvant therapy, post-operative complication, anastomotic leakage classification, Clavien-Dindo classification will be derived from the medical file.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Geraerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided